CLINICAL TRIAL: NCT07300735
Title: A Comparative Study of Diosmin-Hesperidin and Loratadine for the Prevention of G-CSF Induced Bone Pain in Patients With Hematological Malignancies
Brief Title: Comparing Diosmin-Hesperidin and Loratadine to Prevent Bone Pain From G-CSF in Patients With Blood Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB NO:00012098; Serial Number: 0108746 (Other: Ethics Committee Faculty of Medicine Alexandria University); FWA Number: 00018699 (Other: Ethics Committee Faculty of Medicine Alexandria University)
Record Dates: First submitted 2025-12-01; First posted 2025-12-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy; Neutropenia; Bone Pain
Keywords: Loratadine; Diosmin; Filgrastim; Granulocyte Colony Stimulating Factor; G-CSF Induced Bone Pain; Hesperidin; Flavonoid; Antihistamine; Prophylaxis; Randomized Controlled Trial
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia | interventions — Loratadine

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized, open-label clinical trial comparing four interventions for the prevention of G-CSF-induced bone pain: no specific treatment (control), loratadine, diosmin-hesperidin, and the combination of loratadine and diosmin-hesperidin. Participants will be randomly assigned to one of the four groups and will receive their assigned treatment for 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Participants in this arm will receive standard supportive care for G-CSF-induced bone pain, but will not receive the study interventions (loratadine or diosmin-hesperidin).
- Intervention (Active Comparator): Participants in this arm will receive loratadine 10mg tablets once daily, 30 minutes before filgrastim administration, for 5 days.
  Interventions: Drug: Loratadine
- Diosmin-Hesperidin (Experimental): Participants in this arm will receive diosmin-hesperidin 500mg tablets twice daily, 30 minutes before filgrastim administration, for 5 days.
  Interventions: Drug: Diosmin-Hesperidin
- Loratadine + Diosmin-Hesperidin (Experimental): Participants in this arm will receive loratadine 10mg tablets once daily plus diosmin-hesperidin 500mg tablets twice daily, 30 minutes before filgrastim administration, for 5 days.
  Interventions: Drug: Loratadine + Diosmin-Hesperidin

INTERVENTIONS:
Drug: Loratadine — Loratadine 10 mg oral tablet administered once daily, starting 30 minutes before filgrastim administration and continued for 5 consecutive days.
  Arms: Intervention
Drug: Diosmin-Hesperidin — Diosmin-Hesperidin 500 mg oral tablet administered twice daily, starting 30 minutes before daily filgrastim administration and continued for 5 consecutive days.
  Arms: Diosmin-Hesperidin
Drug: Loratadine + Diosmin-Hesperidin — Combination of Loratadine 10 mg oral tablet once daily plus Diosmin-Hesperidin 500 mg oral tablet twice daily, starting 30 minutes before daily filgrastim administration and continued for 5 consecutive days.
  Arms: Loratadine + Diosmin-Hesperidin

SUMMARY:
This is a comparative interventional study to determine the best way to prevent G-CSF induced bone pain in patients with hematological malignancies (blood cancers). G-CSF (Granulocyte Colony-Stimulating Factor) is a drug commonly used in these patients to boost white blood cell production, but it frequently causes severe bone pain.

The study is comparing two oral medications for their effectiveness as a preventive treatment:

* Diosmin-Hesperidin (a flavonoid supplement).
* Loratadine (a common anti-allergy medication).

The core question the study is trying to answer is:

* Is diosmin-hesperidin effective in preventing G-CSF-induced bone pain compared to loratadine?
* Does the combination of diosmin-hesperidin and loratadine offer better pain prevention than either drug alone?

DETAILED DESCRIPTION:
This is a prospective, controlled, randomized, and open-label clinical trial conducted at Alexandria University Hospitals to compare the efficacy of diosmin-hesperidin versus loratadine, and their combination, for the prevention of G-CSF-induced bone pain in adult patients (18-65 years) with hematological malignancies (leukemia or lymphoma) receiving filgrastim.

Rationale:

G-CSF-induced bone pain is a common and debilitating side effect, impacting patient quality of life. While current management strategies using NSAIDs and antihistamines are not always sufficient, diosmin, a flavonoid with known anti-inflammatory and neuroprotective properties, has not been thoroughly investigated for this indication. This study aims to address this gap and explore the potential of diosmin, loratadine, and their combination to mitigate G-CSF-induced bone pain.

Study Design:

Participants meeting the eligibility criteria (detailed elsewhere) will be randomly assigned to one of four treatment groups:

Control Group: No specific treatment for bone pain. Loratadine Group: Loratadine 10mg tablet once daily, administered 30 minutes before filgrastim and continued for 5 days.

Diosmin-Hesperidin Group: Diosmin-Hesperidin 500mg tablet twice daily, administered 30 minutes before filgrastim and continued for 5 days.

Combination Group: Loratadine 10mg tablet once daily plus Diosmin-Hesperidin 500mg tablet twice daily, administered 30 minutes before filgrastim and continued for 5 days.

Filgrastim will be administered according to standard clinical practice for the underlying hematological condition.

Assessments:

Baseline Assessment: Before the start of filgrastim administration, demographic data, medical history (including type of malignancy, comorbidities, prior G-CSF treatment, and chemotherapy details), baseline laboratory tests (CBC, CRP, liver and kidney function), and baseline pain assessment using the Brief Pain Inventory (BPI) will be collected.

Follow-up Assessments:

Within 24 hours of the first filgrastim dose, pain will be assessed using the BPI, and baseline TNF-alpha levels will be measured.

After 5 days of treatment, follow-up laboratory tests (including TNF-alpha levels) and pain assessment using the BPI will be conducted.

Primary Outcome:

The primary outcome is to compare the effectiveness of diosmin-hesperidin, loratadine, and their combination in preventing G-CSF-induced bone pain. This will be assessed by changes in pain frequency and severity (measured by the BPI) and changes in serum TNF-alpha levels.

Secondary Outcome:

The secondary outcome is to identify risk factors associated with the frequency and severity of G-CSF-induced bone pain.

Statistical Analysis:

Data will be analyzed using IBM SPSS version 26. Appropriate statistical tests will be used to compare the treatment groups and assess the relationships between variables.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki and will be subject to approval by the Ethics Committee of Alexandria University. All participants will provide written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years old
* Receiving a G-CSF for one of the following indications:

Treatment of neutropenia along with treatment for leukemia or lymphoma Neutropenia prevention following autologous hematopoietic cell transplant

* Patients with or without bone pain associated with G-CSF administration.
* Willingness to provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with solid tumors.
* Pregnant or breastfeeding women.
* Patients with known allergies or hypersensitivity to Loratadine, Diosmin- Hespiridin or Filgrastim.
* Patients with pre-existing bone disorders or receiving bone modifying agents
* Chronic use of antihistamines, Diosmin-Hespiridin, NSAIDs, corticosteroids, or immunosuppressants.
* Receiving medications with drug interaction grade X with Loratadine, Diosmin-Hespiridin or Filgrastim
* Patients who are unable to understand or provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Bone Pain Severity (Brief Pain Inventory) | Baseline (before first dose of Filgrastim), 24 hours after first Filgrastim dose, and 5 days after treatment initiation.
  This will be measured using the validated Brief Pain Inventory (BPI), which assesses pain intensity (e.g., worst pain, average pain). BPI pain severity will be compared for each trial arm. BPI pain severity will be compared as a composite score (sum of individual pain values divided by 4).
  A score ranging from 0 (no pain) to 10 (worst pain imaginable).
Bone Pain Interference (Brief Pain Inventory) | Baseline (before first dose of Filgrastim), 24 hours after first Filgrastim dose, and 5 days after treatment initiation.
  This will be measured using the validated Brief Pain Inventory (BPI), which assesses the degree to which pain interferes with daily life. BPI pain Interference will be compared for each trial arm. BPI pain interference will be compared as a composite score (sum of individual pain interference values divided by 7).
  A scale of 0 (does not interfere) to 10 (completely interferes).
Change in Serum Tumor Necrosis Factor-alpha (TNF-alpha) Levels | 24 hours after first Filgrastim dose, and After 5 days of the intervention period
  Serum TNF-alpha (pg/mL) is an inflammatory cytokine level measured in the blood that is hypothesized to be elevated in G-CSF induced bone pain. The change from baseline levels will be compared across the four study arms to determine the biological effect of the interventions. Lower levels of TNF-alpha are indicative of a reduction in the inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Moustafa Helmy, Professor, Principal Investigator — Alexandria University; Omar Mohamed Ghallab, Professor, Principal Investigator — Alexandria University; Reham AbdelHalem Abo Elwafa, Professor, Principal Investigator — Alexandria University; Noha Alaa Eldin Hamdy, Assistant professor, Principal Investigator — Alexandria University; Mayssaa Mohamed Elsayed, pharmD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided